CLINICAL TRIAL: NCT05464732
Title: Visual Outcomes, Patient Satisfaction and Spectacle Independence Evaluation of the Acrysof® IQ Vivity® Intraocular Lens Targeted for Emmetropia or Nanovision.
Brief Title: Vivity IOL: Emmetropia Compared to Monovision.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolina Eyecare Physicians, LLC (Other)
Collaborators: Science in Vision (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CEP 20-002
Record Dates: First submitted 2022-07-18; First posted 2022-07-19 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: Patients all had same treatment, evaluated postoperatively in two scenarios.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Monovision then emmetropia (Experimental): The target refraction is plano (0.00 D) for the dominant eye and between -0.50 D and -0.75 D for the non-dominant eye. The Vivity IOL will be implanted bilaterally.
  Corrected vision will involve correcting the dominant eye for emmetropia and the non-dominant eye for -0.50 D.
  Interventions: Device: Vivity IOL emmetropia; Device: Vivity IOL monovision
- Emmetropia then monovision (Experimental): Subject's vision will be tested with both eyes corrected for emmetropia. Subjects will then be tested correcting the dominant eye for emmetropia and the non-dominant eye for -0.50 D.
  Interventions: Device: Vivity IOL emmetropia; Device: Vivity IOL monovision

INTERVENTIONS:
Device: Vivity IOL emmetropia — The Vivity IOL will be implanted bilaterally in all subjects, tested with correction to bilateral emmetropia.
Device: Vivity IOL monovision — The Vivity IOL will be implanted bilaterally in all subjects, tested with correction to emmetropia in the dominant eye and -0.50 in the non-dominant eye.

SUMMARY:
Current visual outcomes expectations of cataract patients are similar to those of refractive surgery patients. Their desire is to be spectacle independent for far, intermediate and near vision activities. Different options are available including: mono-vision and presbyopia correcting intraocular lenses (IOL). Presbyopia correcting IOLs include accommodative, multifocal, trifocal and extended depth of focus (EDOF) IOLs. The Vivity Extended Vision IOL is not a multifocal IOL but due to its design, it provides better intermediate and near VA compared to a monofocal IOL.

DETAILED DESCRIPTION:
The study is concerned with the visual performance of the Vivity Extended Vision IOL at distance, intermediate and near when one of the eyes is targeted for emmetropia and the other is targeted for slight myopia. Patients will serve as their own controls with visual performance evaluated against corrected vision with a target of emmetropia in both eyes.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill the following conditions to qualify for enrollment into the trial

1. Subject is undergoing bilateral lens extraction with intraocular lens implantation.
2. Gender: Males and Females.
3. Age: 50 years and older.
4. Willing and able to provide written informed consent for participation in the study
5. Willing and able to comply with scheduled visits and other study procedures.
6. Scheduled to undergo standard cataract surgery with topical anesthesia in both eyes within 6 to 30 days between surgeries
7. Subjects who require an IOL power in the range of +15.0 D to +25.0 D only.
8. Subjects who require a toric IOL up to +3.00 D at the IOL plane (2.06 D corneal plane).
9. Potential postoperative visual acuity of 0.2 logMAR (20/32 Snellen) or better in both eyes.

Exclusion Criteria:

Subjects with any of the following conditions on the eligibility exam may not be enrolled into the trial.

1. Severe preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, retinal detachment, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmos or macrophthalmos, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc.
2. Uncontrolled diabetes.
3. Use of any systemic or topical drug known to interfere with visual performance.
4. Contact lens use during the active treatment portion of the trial.
5. Any concurrent infectious/non-infectious conjunctivitis, keratitis or uveitis.
6. Clinically significant corneal dystrophy
7. History of chronic intraocular inflammation.
8. History of retinal detachment.
9. Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
10. Previous intraocular surgery.
11. Previous corneal refractive surgery (i.e. laser-assisted in situ keratomileusis, photorefractive keratectomy, radial keratotomy).
12. Previous keratoplasty
13. Severe dry eye
14. Pupil abnormalities
15. Anesthesia other than topical anesthesia (i.e. retrobulbar, general, etc).
16. Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
17. Participation in (or current participation) any ophthalmic investigational drug or ophthalmic device trial within the previous 30 days prior to the start date of this trial.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates the patient is unsuitable for the trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Solomon, Principal Investigator — Carolina Eyecare Physicians, LLC
Locations (1):
- Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 33 subjects were enrolled in the study. One was lost to follow up and one experienced a progression of their macular degeneration, leaving 31 subjects for analysis.
Groups:
- Monovision Then Emmetropia; Emmetropia Then Monovision: All study participants received the Vivity IOL in both eyes.
  1. Target refraction plano (emmetropia): the target was (0.00 D) for both the dominant and the non-dominant eye. Corrected vision will involve correcting both eyes for plano.
  2. Target refraction monovision where the target was (0.00 D) for the dominant eye and between -0.50 D and -0.75 D for the non-dominant eye. Corrected vision will involve correcting the dominant eye for emmetropia and the non-dominant eye for -0.50 D.
Period: Overall Study
Arm/Group | Monovision Then Emmetropia | Emmetropia Then Monovision
Started | 16 | 17
Completed | 15 | 16
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: All study participants received the Vivity IOL in both eyes.
  The same group of participants were evaluated twice using two different target refractions:
  1. Target refraction plano: the target was (0.00 D) for both the dominant and the non-dominant eye. Corrected vision will involve correcting both eyes for plano.
  2. Target refraction monovision where the target was (0.00 D) for the dominant eye and between -0.50 D and -0.75 D for the non-dominant eye. Corrected vision will involve correcting the dominant eye for emmetropia and the non-dominant eye for -0.50 D.
  Participants were randomized to which target was evaluated first and there was a 10 minutes break between the 2 evaluations.
Arm/Group | Overall
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Binocular Uncorrected Near (40 cm) Visual Acuity
Description: The logMAR binocular uncorrected visual acuity at 40 cm will be measured.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Monovision: The target refraction is plano (0.00 D) for the dominant eye and between -0.50 D and -0.75 D for the non-dominant eye. The Vivity IOL will be implanted bilaterally.
  Corrected vision will involve correcting the dominant eye for emmetropia and the non-dominant eye for -0.50 D.
  Vivity IOL: The Vivity IOL will be implanted bilaterally in all subjects.
- Emmetropia: Subject's vision will be tested with both eyes corrected for emmetropia.
  Vivity IOL: The Vivity IOL will be implanted bilaterally in all subjects.
Arm/Group | Monovision | Emmetropia
Number analyzed (Participants) | 31 | 31
logMAR | 0.21 (0.11) | 0.39 (0.16)

ADVERSE EVENTS:
Time Frame: 3 months
Description: AE were collected from the time the ICF was signed to the exit visit at 3 months.
Arm/Group | Monovision | Emmetropia
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT05464732/Prot_SAP_000.pdf